CLINICAL TRIAL: NCT03564483
Title: Prospective Registry of Gynecologic Patients With Extramammary Paget's Disease
Brief Title: Gynecologic Extramammary Paget's Disease
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 17-007532
Record Dates: First submitted 2018-06-11; First posted 2018-06-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Extramammary Paget's Disease; Extramammary Paget Disease; Paget Disease, Extramammary; Extramammary Paget's Disease of Vulva (Diagnosis); Extramammary Paget's Disease of Vagina (Diagnosis); Extramammary Paget's Disease Vulva Invasive; Extramammary Paget's Disease of Anus (Diagnosis); Extramammary Paget's Disease of Anal Canal (Diagnosis); Extramammary Paget's Disease of Skin
MeSH Terms: conditions — Paget Disease, Extramammary; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissues will be obtained in order to perform tumor molecular profiling to identify targetable somatic mutations in EMPD.
  The vulvar and perianal microbiome of women with extramammary Paget's disease will be evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Registry Observational Study: All women presenting for evaluation of Extramammary Paget's Disease (EMPD) at Mayo Clinic in Rochester MN.

SUMMARY:
In addition to evaluating treatment outcomes, tissue samples and swabs will be collected as part of this study to allow physicians to better understand Extramammary Paget's Disease (EMPD). The researchers also want to learn more about the microorganisms (microbiome) that live on or near the areas of skin affected by EMPD, in order to better understand this condition.

DETAILED DESCRIPTION:
This is a prospective cohort study. Patients with Extramammary Paget's Disease (EMPD), specifically women with vulvar/perianal Paget's disease, will be identified during presentation to either the Dermatology Department or Gynecologic Surgery department at Mayo Clinic.

During physical exam, the patients will undergo skin/rectum/vagina cultures to evaluate the microbiome in these patients. The patients will be entered into the established care pathway for EMPD. They will be asked to complete sexual health questionnaires including: The Women's Health Clinical Questionnaires include the Menopause Rating Scale (MRS)1, Perceived Stress Scale2, Brief Resilience Scale (BRS)3, LASA Quality of Life Assessment4, Female Sexual Function Index (FSFI)5, Female Sexual Distress Scale-Revised6, Kansas Marital Satisfaction Scale7, and Pittsburgh Sleep Quality Index (PSQI)8.

The patients will be referred to Women's Health Clinic as part of the care pathway and will undergo preoperative genital sensory testing (GST) which measures sensation of the clitoris, vulva, and vagina. The patients will have a Dermatology consultation and Moh's micrographic procedure as indicated. If choosing to proceed with surgical intervention, the patients will then undergo an excisional procedure with the Department of Gynecologic surgery. Swabs, urine and tissue will be collected prior to procedures or surgery for microbiome analysis.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Age 18 years or older
* Diagnosed with primary or recurrent EMPD of vulva and/or perianal region of the body
* Willing and able to provide signed informed consent

Exclusion Criteria:

* Males
* Diagnosis of Paget's Disease in body areas other than vulvar or perianal region

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with Extramammary Paget's Disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02-19 (Actual); Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Collect prospective data including outcomes and long-term survival in women with extramammary Paget's disease (EMPD). | 25 years
  Prospective data including patient demographic information, surgical outcomes, surgical morbidity, recurrence, and long-term survival in extramammary Paget's disease (EMPD) will be collected as part of this registry..

CONTACTS AND LOCATIONS:
Overall Officials: Jamie N. Bakkum-Gamez, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruce KH, Kilts TP, Lohman ME, Vidal NY, Fought AJ, McGree ME, Keeney GL, Baum CL, Brewer JD, Bakkum-Gamez JN, Cliby WA. Mohs surgery for female genital Paget's disease: a prospective observational trial. Am J Obstet Gynecol. 2023 Dec;229(6):660.e1-660.e8. doi: 10.1016/j.ajog.2023.08.018. Epub 2023 Aug 24. PMID 37633576